CLINICAL TRIAL: NCT05821933
Title: An Open Single-arm Study to Evaluate the Safety, Tolerability, Efficacy of RC108 in Combination With Furmonertinib and Toripalimab in Patients With Advanced EGFR-mutated NSCLC Ib/II Study
Brief Title: RC108 Combine With Furmonertinib With/Without Toripalimab in Patients With EGFR-mutated NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC108-C003
Record Dates: First submitted 2023-03-13; First posted 2023-04-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: NSCLC
MeSH Terms: interventions — aflutinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1 RC108 plus Furmonertinib (Experimental): phaes 1: RC108 plus Furmonertinib
  Interventions: Drug: RC108
- cohort 2 RC108 plus Furmonertinib and Toripalimab (Experimental): phaes 1: RC108 plus Furmonertinib and Toripalimab
  Interventions: Drug: RC108
- cohort 3 RP2D RC108 plus Furmonertinib (Experimental): phaes 2: RP2D RC108 plus Furmonertinib
  Interventions: Drug: RC108
- cohort 4 RP2D RC108 plus Furmonertinib and Toripalimab (Experimental): phaes 2: RP2D RC108 plus Furmonertinib and Toripalimab
  Interventions: Drug: RC108

INTERVENTIONS:
Drug: RC108 — RC108 plus Furmonertinib and/or Toripalimab
  Other Names: Furmonertinib; Toripalimab

SUMMARY:
an open, single-arm, multicenter phase Ib/II study

DETAILED DESCRIPTION:
an open, single-arm, multicenter phase Ib/II study evaluated the safety, tolerability, efficacy and pharmacokinetic profile of RC108 in combination with Furmonertinib or in combination with Furmonertinib and Toripalimab in patients with locally advanced or metastatic EGFR MET-expressing mutated NSCLC who have failed EGFR-TKI, and to develop a reasonable follow-up study for combination dosing regimens

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign an informed consent form.
2. Age between 18 and 75 years old (inclusive).
3. Expected survival period of at least 12 weeks as determined by the investigator.
4. ECOG performance status of 0 or 1.
5. For female subjects: must be surgically sterile, postmenopausal, or willing to use a medically accepted contraceptive method (such as an intrauterine device, birth control pills, or condoms) during the study treatment period and for 6 months after the end of the study treatment. A negative pregnancy test within 7 days before study treatment initiation is required, and the subject must not be breastfeeding. For male subjects: must be surgically sterile or willing to use a medically accepted contraceptive method during the study treatment period and for 6 months after the end of the study treatment.
6. Able to understand the trial requirements, willing and able to comply with trial and follow-up procedures.
7. Bone marrow function:

   Hemoglobin ≥9 g/dL Absolute neutrophil count (ANC) ≥1.5 × 10^9/L Platelet count ≥100 × 10^9/L
8. Liver function (based on the clinical trial center's normal values):

   Serum total bilirubin ≤1.5 times the upper limit of normal (ULN) ALT and AST ≤2.5 × ULN and serum total bilirubin ≤1.5 times the ULN if there is no liver metastasis; ALT and AST ≤5 × ULN and serum total bilirubin ≤2 times the ULN if there is liver metastasis.
9. Kidney function (based on the clinical trial center's normal values):

   Serum creatinine ≤1.5 × ULN, or calculated creatinine clearance (CrCl) by the Cockcroft-Gault formula ≥60 mL/min, or measured 24-hour urine CrCl ≥60 mL/min.
10. Heart function:

    NYHA class <3 Left ventricular ejection fraction (LVEF) ≥50% QTc interval ≤450 ms
11. All subjects must have locally advanced or metastatic non-small cell lung cancer (NSCLC) confirmed by histology or cytology.
12. Must have at least one EGFR-sensitive mutation: exon 19 deletion, L858R mutation in exon 21, T790M mutation in exon 20, G719X mutation in exon 18, S768I mutation in exon 20, or L871Q mutation in exon 21 (inclusion of patients with exon 20 insertion mutation is allowed).
13. Must have received approved first/second/third-generation EGFR-TKI treatment in the past and experienced radiological progression during EGFR-TKI treatment. The patient is allowed to have received other systemic treatments such as chemotherapy and anti-angiogenic agents, regardless of the sequence with EGFR-TKI treatment.
14. Must provide a tumor tissue sample that meets the central laboratory's testing requirements and has MET (IHC) expression of 1+, 2+, or 3+ as determined by the central laboratory.
15. Must agree to provide tumor tissue or blood samples collected during or after previous EGFR-TKI treatment-induced radiological progression for EGFR T790M detection or provide the results of EGFR T790M detection in the tumor tissue sample.
16. Must provide the most recent tumor tissue sample for PD-L1 expression testing, which will be used to stratify subjects for randomization.
17. At least one measurable lesion according to RECIST 1.1 criteria.

Exclusion Criteria:

1. Have used an investigational drug within 4 weeks prior to the start of study dosing.
2. Have undergone major surgery within 4 weeks prior to the start of study dosing and have not fully recovered.
3. Received a live vaccine within 4 weeks prior to the start of study dosing or are scheduled to receive any vaccine (except novel inactivated coronavirus vaccine) during the study period.
4. An arterial/venous thrombotic event such as a cardiovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism within 6 months prior to study dosing.
5. Clinically significant QT interval prolongation or other arrhythmias or clinical states that, in the opinion of the investigator, have the potential to increase the risk of QT interval prolongation; e.g., resting state ECG QTc > 450 ms, complete left bundle branch block, third degree AV block, congenital long QT syndrome, severe hypokalemia, or ongoing medication that can cause QT interval prolongation.
6. The presence of preexisting or ongoing interstitial lung disease (ILD), drug-induced interstitial lung disease, radiation pneumonia requiring steroid medication, or those with clinical manifestations of suspected interstitial lung disease.
7. The presence of clinically uncontrollable third interstitial fluid, such as pleural effusion, peritoneal effusion, or pericardial effusion that is clinically symptomatic and cannot be controlled by drainage or other means and is, in the judgment of the investigator, unenrollable.
8. Suffering from systemic diseases that are not under stable control, including diabetes, hypertension, pulmonary fibrosis, acute and chronic lung disease, interstitial lung disease, cirrhosis of the liver, etc.
9. Known to have a psychiatric or substance abuse disorder that may have an impact on compliance with trial requirements
10. Ongoing active infection requiring systemic treatment, such as severe pneumonia, sepsis, etc.
11. The presence or suspicion of active tuberculosis.
12. Known presence and activity of any of the following infectious diseases: positive HIV antibody test result; positive HBsAg with positive HBV DNA (i.e., copy number ≥ 2000 copies/ml); positive HCV antibody with positive HCV RNA.
13. Those who have used a strong inhibitor of cytochrome P450 3A4 (CYP3A4) within 7 days prior to the first dose or a strong inducer of CYP3A4 within 21 days
14. Have any other disease, metabolic abnormality, physical examination abnormality, or laboratory test abnormality that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that is inappropriate for the use of the study drug, or that will affect the interpretation of the study results, or that places the patient at high risk
15. Women who are pregnant or breastfeeding or women/men who are planning to have children.
16. Subjects who are estimated to have insufficient patient compliance to participate in this clinical study or who, in the opinion of the investigator, have other factors that make them inappropriate for participation in this study.
17. Known small cell lung cancer transformation or the presence of a small cell component.
18. Presence of brain metastases and/or cancerous meningitis. Subjects who have been treated for brain metastases may be considered for participation in this study provided that the disease has been stable for at least 3 months, no disease progression has occurred as determined by imaging within 4 weeks prior to the first dose of study treatment, all neurological symptoms have returned to baseline levels, there is no evidence of new or expanding brain metastases, and treatment with radiation, surgery, or steroids has been discontinued at least 28 days prior to the first dose of study treatment . This exception does not include meningeal metastases and carcinomatous meningitis, which should be excluded regardless of their clinical stability.
19. Other malignancies (except non-melanoma skin cancer, cervical carcinoma in situ or other tumors that have been effectively treated and are considered cured) within 5 years prior to signing the informed consent form.
20. Known hypersensitivity or delayed allergic reactions to certain components of RC108 for injection, vomitinib or similar drugs, in addition to non-enrollment in Cohort 2 and Cohort 4 for hypersensitivity or delayed allergic reactions to certain components of treprolizumab or similar drugs
21. Have received drugs targeting the HGF and/or MET pathways prior to study administration.
22. Prior use of PD-1/L1 inhibitors is inadmissible to Cohort 2 and Cohort 4.
23. Chemotherapy, radiotherapy, immunotherapy and targeted therapy received prior to the start of study dosing less than 4 weeks or less than 5 half-lives (whichever is shorter) from the first dose of this study.
24. Hormonal therapy received within 2 weeks prior to the start of study dosing for the tumor(s) affected.
25. Received palliative radiotherapy targeting bone metastases within 2 weeks prior to the start of study dosing.
26. Having received antitumor herbal therapy within 2 weeks prior to the start of study dosing
27. Toxicity of prior antitumor therapy that have not recovered to CTCAE [version 5.0] grade 0-1, with the following exceptions: a. alopecia; b. hyperpigmentation; c. long-term toxicity due to radiotherapy that, in the judgment of the investigator, cannot be recovered.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Dose limiting toxicity (DLT) | 21-days
  To observe the durability and safety of RC108 plus Furmonertinib or plus Furmonertinib and Toripalimab in patients with advanced after single and multiple administration, observe the dose limiting toxicity (DLT)and the reversibility of toxicity

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months
  Tumor response was assessed by investigator according to RECIST v1.1
Duration of Response (DOR) | up to 24 months
  DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier
Disease control rate (DCR) | up to 24 months
  DCR was defined as the proportion of patients who achieved an objective response or maintained stable disease during the study
Overall Survival(OS) | up to 24 months
  OS was defined as the time from the first study treatment to the date of death from any cause
Maximum tolerated dose (MTD) | 21-days
  To observe the durability and safety of RC108 plus Furmonertinib or plus Furmonertinib and Toripalimab in patients with advanced after single and multiple administration, observe the maximum tolerated dose (MTD)，the relationship between toxicity and dose

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China